CLINICAL TRIAL: NCT04887064
Title: An Open-label Single-dose Study to Evaluate the Pharmacokinetics of Sotorasib in Healthy Subjects and Subjects With Moderate or Severe Hepatic Impairment
Brief Title: Pharmacokinetics of Sotorasib in Healthy Participants and Participants With Moderate or Severe Hepatic Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 20200362
Expanded Access: NCT04667234 (No longer available)
Record Dates: First submitted 2021-05-11; First posted 2021-05-14 (Actual); Results first posted 2024-04-19 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2023-01

CONDITIONS: Hepatic Impairment
Keywords: Hepatic Impairment; Sotorasib
MeSH Terms: interventions — sotorasib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Normal Hepatic Function (Experimental)
  Interventions: Drug: Sotorasib
- Moderate Hepatic Impairment (Experimental)
  Interventions: Drug: Sotorasib
- Severe Hepatic Impairment (Experimental)
  Interventions: Drug: Sotorasib

INTERVENTIONS:
Drug: Sotorasib — Sotorasib will be administered as an oral tablet.
  Other Names: AMG 510

SUMMARY:
The main purpose of the study is to evaluate the pharmacokinetics (PK) of a single oral dose of sotorasib administered in participants with moderate or severe hepatic impairment compared to participants with normal hepatic function.

ELIGIBILITY:
Key Inclusion Criteria

All Participants

* Participant has provided informed consent before initiation of any study-specific activities/procedures
* Participants between 18 and 70 years of age
* Body mass index between 18 and 38 kg/m^2
* Females of nonchildbearing potential defined as permanently sterile or postmenopausal

Participants with Normal Hepatic Function

* In good health, determined by no clinically significant findings from medical history, physical examination, 12-lead ECG, vital signs measurements, and clinical laboratory evaluations

Participants with Hepatic Impairment

* Child-Pugh B or C classification with clinical laboratory values and clinical examination findings
* Documented medical history of chronic liver disease

Key Exclusion Criteria

All Participants

* Female participants with a positive pregnancy test at Screening or Check-in
* Male participants with a pregnant partner or partner planning to become pregnant who are unwilling to practice abstinence or use a condom for 7 days after dosing
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance
* Participant has received a dose of an investigational drug (new chemical entity) within the past 30 days or 5 half-lives, whichever is longer, prior to Check-in
* Use of any over-the-counter or prescription medications within 30 days or 5 half-lives (whichever is longer)
* All herbal medicines vitamins, and supplements consumed by the subject within the 30 days prior to enrollment
* Alcohol consumption from 48 hours prior to Check-in
* Positive test for illicit drugs, cotinine (tobacco or nicotine use), and/or alcohol use at Check-in
* Positive human immunodeficiency virus test at Screening

Participants with Normal Hepatic Function

* Positive hepatitis B or hepatitis C panel at Screening. Subjects whose results are compatible with prior immunity (vaccination or prior infection) may be included
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > upper limit of normal (ULN) at Screening or Check-in
* Total bilirubin levels > ULN at Screening or Check-in
* A QT interval corrected for heart rate based on the Fridericia correction (QTcF) interval > 450 msec in male subjects or > 470 msec in female subjects or history/evidence of long QT syndrome at Screening or Check-in, confirmed by calculating the mean of the original value and 2 repeats

Participants with Hepatic Impairment

* Values outside the normal range for liver function tests that are not consistent with their hepatic condition, as determined by the Investigator (or designee)
* A QTcF interval > 470 msec in male subjects or > 480 msec in female subjects at Screening or Check-in, confirmed by calculating the mean of the original value and 2 repeats
* Use of a new medication, or a change in dose, for the treatment, or worsening of, hepatic encephalopathy within 30 days prior to Check-in
* Presence of a portosystemic shunt
* Evidence of severe ascites

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-04-22 (Actual); Primary Completion 2022-03-09 (Actual); Study Completion 2022-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (5):
- United States (5):
  - Orange County Research Center, Tustin, California
  - Clinical Pharmacology Of Miami LLC, Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida
  - American Research Corporation, San Antonio, Texas
  - Pinnacle Clinical Research - San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at research centers in the United States from April 2021 to March 2022.
Groups:
- Normal Hepatic Function: Participants with normal hepatic function (no impairment) received a single oral 960 mg dose of sotorasib under fasted conditions.
- Moderate Hepatic Impairment: Participants with moderate hepatic function (Child-Pugh Class B at screening) received a single oral 960 mg dose of sotorasib under fasted conditions.
- Severe Hepatic Impairment: Participants with severe hepatic function (Child-Pugh Class C at screening) received a single oral 960 mg dose of sotorasib under fasted conditions.
Period: Overall Study
Arm/Group | Normal Hepatic Function | Moderate Hepatic Impairment | Severe Hepatic Impairment
Started | 7 | 8 | 5
Completed | 7 | 8 | 5
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population: All participants who received sotorasib and had at least 1 postdose safety assessment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Normal Hepatic Function | Moderate Hepatic Impairment | Severe Hepatic Impairment | Total
Number analyzed (Participants) | 7 | 8 | 5 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.0 (7.35) | 58.5 (5.66) | 51.6 (7.37) | 57.0 (7.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 2 | 9
  Male | 4 | 4 | 3 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 6 | 3 | 13
  Not Hispanic or Latino | 3 | 2 | 2 | 7
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 6 | 8 | 4 | 18
  Black or African American | 1 | 0 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Sotorasib
Time Frame: Predose (Hour 0), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120, 144, and 168 hours postdose following administration of sotorasib on Day 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Normal Hepatic Function | Moderate Hepatic Impairment | Severe Hepatic Impairment
Number analyzed (Participants) | 7 | 8 | 5
ng/mL | 5080 (108.5) | 4850 (60.6) | 7250 (15.7)

2. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to the Last Quantifiable Concentration (AUClast) of Sotorasib
Time Frame: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Normal Hepatic Function | Moderate Hepatic Impairment | Severe Hepatic Impairment
Number analyzed (Participants) | 7 | 8 | 5
h*ng/mL | 28700 (87.8) | 21500 (58.2) | 29900 (12.6)

3. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to Infinity (AUCinf) of Sotorasib
Time Frame: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Normal Hepatic Function | Moderate Hepatic Impairment | Severe Hepatic Impairment
Number analyzed (Participants) | 7 | 8 | 5
h*ng/mL | 29000 (86.4) | 21700 (58.2) | 30100 (12.2)

4. Secondary Outcome: Number of Participants Who Experienced One or More Treatment Emergent Adverse Events (TEAEs)
Description: TEAEs were defined as any adverse events (AEs) that started during or after dosing, or started prior to dosing and increased in severity after dosing.
  Any clinically significant changes in clinical laboratory evaluations, 12-lead electrocardiograms (ECGs) and vital signs were also reported as TEAEs.
Time Frame: Day 1 to Day 8
Measure: Count of Participants; unit: Participants
Arm/Group | Normal Hepatic Function | Moderate Hepatic Impairment | Severe Hepatic Impairment
Number analyzed (Participants) | 7 | 8 | 5
Participants | 1 | 2 | 1

5. Secondary Outcome: Unbound Cmax (Cmax,u) of Sotorasib
Time Frame: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Normal Hepatic Function | Moderate Hepatic Impairment | Severe Hepatic Impairment
Number analyzed (Participants) | 7 | 8 | 5
ng/mL | 183 (240.8) | 400 (110.9) | 1220 (9.8)

6. Secondary Outcome: Unbound AUClast (AUClast,u) of Sotorasib
Time Frame: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Normal Hepatic Function | Moderate Hepatic Impairment | Severe Hepatic Impairment
Number analyzed (Participants) | 7 | 8 | 5
h*ng/mL | 694 (146.3) | 1320 (71.0) | 4680 (29.4)

7. Secondary Outcome: Unbound AUCinf (AUCinf,u) of Sotorasib
Time Frame: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Normal Hepatic Function | Moderate Hepatic Impairment | Severe Hepatic Impairment
Number analyzed (Participants) | 7 | 8 | 5
h*ng/mL | 742 (156.7) | 1340 (69.6) | 4680 (29.4)

8. Secondary Outcome: Unbound Apparent Total Plasma Clearance (CLu/F) of Sotorasib
Time Frame: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Normal Hepatic Function | Moderate Hepatic Impairment | Severe Hepatic Impairment
Number analyzed (Participants) | 7 | 8 | 5
L/h | 1290 (156.7) | 715 (69.6) | 205 (29.4)

9. Secondary Outcome: Unbound Apparent Volume of Distribution During the Terminal Phase (Vz,u/F) of Sotorasib
Time Frame: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | Normal Hepatic Function | Moderate Hepatic Impairment | Severe Hepatic Impairment
Number analyzed (Participants) | 7 | 8 | 5
liters | 7080 (275.6) | 3820 (115.2) | 928 (39.1)

ADVERSE EVENTS:
Time Frame: Day 1 to Day 8
Description: All participants who received 960 mg single oral dose of sotorasib, including participants with no hepatic impairment, moderate hepatic impairment and severe hepatic impairment.
Groups:
- Normal Hepatic Function: Normal Hepatic Function
- Moderate Hepatic Impairment: Moderate Hepatic Impairment
- Severe Hepatic Impairment: Severe Hepatic Impairment
Arm/Group | Normal Hepatic Function | Moderate Hepatic Impairment | Severe Hepatic Impairment
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/8 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/8 | 0/5
Other Adverse Events (participants affected / at risk) | 1/7 | 2/8 | 1/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Normal Hepatic Function (N=7) | Moderate Hepatic Impairment (N=8) | Severe Hepatic Impairment (N=5)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram qt prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1)
Sensory disturbance (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2021-02-09): https://cdn.clinicaltrials.gov/large-docs/64/NCT04887064/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-02): https://cdn.clinicaltrials.gov/large-docs/64/NCT04887064/SAP_001.pdf